CLINICAL TRIAL: NCT06303323
Title: Comparative Effectiveness of Qigong Exercise Versus Wu Dang Tai Chi Chuan on Exercise Capacity and Stress in CVD Risk Individuals
Brief Title: Comparative Effectiveness of Qigong Exercise Versus Wu Dang Tai Chi Chuan in CVD Risk Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01816 Nawal Fatima
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Diseases; Risk Behavior, Health
Keywords: Qigong exercise; Wu Dang Tai Chi Chuan; Exercise capacity; CVD Risk individuals
MeSH Terms: conditions — Cardiovascular Diseases; Health Risk Behaviors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong Exercise (Experimental): Baduanjin Exercise will be performed which consists of 8 standing postures. At least 30 minutes per time. 10-13 min for a set of Badaunjin
  Interventions: Other: Qigong Exercise
- Wu Dang Tai Chi (Experimental): Wu Dang 13 form postures will be performed. Initially, each posture will be performed 3 times then progressively increase to more according to the patient's discomfort.
  Interventions: Other: Wu Dang Tai Chi

INTERVENTIONS:
Other: Qigong Exercise — Baduanjin Exercise will be performed which consists of 8 standing postures. At least 30 minutes per time. 10-13 min for a set of Badaunjin.
  In the first 2 weeks, two sets of Baduanjin will be performed. Total Duration: 6 weeks Frequency: for 3 days/week. (alternative days) Intensity: low-intensity exercise Total Time: 50 Minutes Type: aerobic training
  Arms: Qigong Exercise
Other: Wu Dang Tai Chi — Wu Dang 13 form postures will be performed. Initially, each posture will be performed 3 times then progressively increase to more according to the patient's discomfort.
  Total Duration: 6 weeks Frequency: 3 times/ week (alternative day ) Intensity: Low to Moderate Intensity Time: 50 Minutes Type: aerobic training
  Arms: Wu Dang Tai Chi

SUMMARY:
To compare whether the Qigong exercise or Wu Dang Tai Chi Chuan will be effective in improving exercise capacity and reducing stress in CVD-risk individuals. Based on preliminary data, Qigong and Tai-Chi may help treat anxiety and depression symptoms in patients with chronic illnesses as well as in healthy adults. Without the need for specialized equipment, Qigong and Tai-Chi are both readily adjustable mind-body exercises that may be done whenever and wherever. For this reason, Qigong and TaiChi should be extensively encouraged as ways to enhance emotional wellbeing

DETAILED DESCRIPTION:
Since no comparison study has thus far been carried out in Pakistan which includes both interventions and very little literature is available. They belong to a group of Chinese exercises known for their efficacy in reducing blood pressure, stress, and quality of life and improving exercise capacity in patients with a high risk of CVD or CVD disease. These techniques are cost-effective treatment approaches and provide early outcomes. The positive results of this study would be helpful in the near future.

ELIGIBILITY:
Inclusion Criteria:

* According to the Framingham risk calculator 10% to 20%+ for moderate to high-risk
* Patients at risk of CVD (last 6 months)
* Patients with either HTN, dyslipidemia, or diabetes
* Patients with less than 45 scores on the Berg Balance scale
* Stress from moderate to severe on PSS
* No regular physical exercise for at least 1 year
* Willing to take part

Exclusion Criteria:

* History of stroke
* CVD
* Acute Infection
* Acute injury
* Any diagnosed psychological issue
* MSK disorders
* Member of marital arts/dance

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 6 weeks
  Changes from baseline to 6 weeks after the intervention, measured through 6 min walk test (6 MWT). It is a submaximal exercise test that can aid in assessing the functional/exercise capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.
Stress | 6 weeks
  Changes from baseline to 6 weeks after the intervention, measured through Perceived Stress Scale.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No